CLINICAL TRIAL: NCT01705795
Title: Anti-IL-5 Therapy in Bullous Pemphigoid. Randomized, Placebo-controlled, Double-blind Study Evaluating the Effect of Anti-IL-5 Therapy in Patients With Bullous Pemphigoid.
Brief Title: Anti-IL-5 Therapy in Bullous Pemphigoid (BP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191/11
Record Dates: First submitted 2012-10-05; First posted 2012-10-12 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Pemphigoid, Bullous
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — mepolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mepolizumab (Active Comparator): Mepolizumab 750 mg four times one month apart.
  Interventions: Drug: Mepolizumab (a-IL-5 antibody)
- Placebo (Placebo Comparator): Placebo (saline) four times one month apart
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mepolizumab (a-IL-5 antibody) — 750mg mepolizumab four times over four months
  Arms: Mepolizumab
Drug: Placebo — Nacl four times over four months
  Arms: Placebo

SUMMARY:
Randomized, placebo-controlled, double-blind study evaluating the effect of anti-IL-5-therapy in patients with bullous pemphigoid. The primary study objective is to determine the efficacy of an anti-IL-5 monoclonal antibody therapy, administered as 750mg mepolizumab, in patients with bullous pemphigoid.

DETAILED DESCRIPTION:
Background

Bullous pemphigoid (BP) is the most common autoimmune blistering skin disease. It characteristically affects the elderly (>70 years) with an annual incidence of 5 to 35 per million. This is comparable with the incidence of eosinophilic esophagitis that we determined with approximately 14 per million. Eosinophilic esophagitis has been recognized as an emerging medical problem and, consequently, several studies with anti-IL-5-antibodies have been performed and are still ongoing. It should be noted, however, that, in contrast to eosinophilic esophagitis, the incidence of BP is dramatically increasing with an average of 17% per year. Moreover, with the increase of the proportion of the elderly in the industrialized world, the medical problems associated with BP will even be more visible in the near future. For instance, patients with BP have an increased mortality risk of 2.3. In the US, an increase in mortality of BP patients has been noticed from 1979 to 2002. Taken together, BP is a frequent disease that affects mostly the elderly.

BP often starts with extremely pruritic skin lesions resembling eczema or urticaria before vesicles and blisters arise. In 10-30% of patients, BP also involves the oral mucosa. Disease severity can be determined by means of the autoimmune bullous skin disorder intensity score (ABSIS) that evaluates the involved area as well as the disease activity. The disease is due to an autoimmune response to structural components of junctional adhesion complexes leading to the damage of the dermal-epidermal junction with subepidermal blister formation. Specifically, autoreactive B and T cell responses against the hemidesmosomal antigens BP180 and BP230 have been identified. Serum levels of autoantibodies to BP180 reflect the disease severity and activity. The T cells are memory CD4+ cells producing both Th1 and Th2 cytokines, mostly IL-4, IL-5 and IL-13. IL-5 as well as eotaxin are abundantly found in blister fluids. The production of IL-5 is indeed associated with blood eosinophilia and significant eosinophil infiltration in the skin of BP patients. Eosinophils are thought to be critically implicated in blister formation by releasing toxic granule proteins (ESP, MBP) and proteolytic enzymes.

Systemic corticosteroids have been widely used for the treatment of BP. Nevertheless, the use of steroids is limited by their side effects. in therapy-resistant cases, immunosuppressive drugs such as azathioprine, chlorambucil, cyclophosphamide, cyclosporine, methotrexate, mycophenolate mofetil are employed, but their corticosteroid-sparing effect and overall benefit in BP is highly disputed. 70% of the relapses are usually observed within three months, 85% within 6 months after stopping therapy.

Since eosinophils are characteristically found in the skin at early stages of the disease before blisters occur and contribute to tissue damage, targeting eosinophils by reducing their number and activation might thus be a promising alternative therapeutic approach. Anti-IL-5 antibody therapy has been shown to be effective in depleting eosinophils, e.g. in diseases such as eosinophilic esophagitis and hypereosinophilic syndrome.

Objective

To determine the safety and efficacy of mepolizumab in patients with bullous pemphigoid.

Methods

clinical trial with 750 mg mepolizumab over three months, evaluate time period from start of therapy until relapse, ABSIS-Score, Pruritus Score, Antibody levels, immuno pathological evaluation of skin biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Men, women >18 years
* Active BP (diagnosed by typical clinical picture and skin biopsy)
* Must give written informed consent

Exclusion Criteria

* Patients with other skin disease
* Patients with severe diseases of other organ systems
* Systemic treatment for BP
* Topical therapy with corticosteroids and other anti-inflammatory substances
* For female patients, unless postmenopausal or surgically sterile, unwillingness to practice effective contraception (defined as methods with <1% failure rate)
* Female patients who are currently pregnant or breast-feeding
* Current abuse of alcohol and/or drugs
* History of or a new diagnosis or treatment of an invasive malignancy within 5 years of enrollment. Patients with a history of treated squamous cell and/or basal cell carcinomas limited to the skin are not excluded.
* History of recurrent clinically significant infection
* Congenital or acquired immunodeficiency syndrome
* Current enrollment in any other investigational drug study
* Previous participation in this study or previous studies with mepolizumab
* Hypersensitivity to mepolizumab or its constituents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-02-13 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Time period (in days) from start of therapy until relapse, mepolizumab vs placebo | Before, at 3-9 months

SECONDARY OUTCOMES:
Changes of BP severity score over time (ABSIS) | At baseline, during therapy (expected to be ca. 4 months), follow up (expected to be ca. 9 months)
Changes of pruritus score (visual analog scale) | At baseline, during therapy (expected to be ca. 4 months), follow up (expected to be ca. 9 months)
Changes of BP-antibody titers over time | At baseline, during therapy (expected to be ca. 4 months), follow up (expected to be ca. 9 months)
Number of patients with AE, severity of AE | At baseline, during therapy (expected to be ca. 4 months), follow up (expected to be ca. 9 months)

CONTACTS AND LOCATIONS:
Overall Officials: Dagmar Simon, Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- Dep. of Dermatology, Bern University Hospital, Bern, Switzerland